CLINICAL TRIAL: NCT05272241
Title: Registry of Asthma Characterization and Recruitment 3 (RACR3) (CAUSE-02)
Brief Title: Registry of Asthma Characterization and Recruitment 3 (RACR3)
Acronym: RACR3
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT CAUSE-02
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Asthma
Keywords: Asthma; Allergy; CAUSE; RACR
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Biospecimen Retention: Samples Without DNA — Whole Blood Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-center, non-interventional registry to create and maintain a database of participants to serve as a recruitment source for current and future DAIT NIAID-sponsored Childhood Asthma in Urban Settings (CAUSE) studies.

DETAILED DESCRIPTION:
Protocol CAUSE-02 RACR3 is a multi-center, non-interventional registry to create and maintain a database of participants to serve as a recruitment source for current and future DAIT NIAID-sponsored Childhood Asthma in Urban Settings (CAUSE) studies. Approximately 1,500 participants - of all ages, living in selected Office of Management and Budget (OMB) defined Metropolitan Statistical Areas (MSAs) will be enrolled in the registry.

The registry database will be generated with data gathered at a single core visit, followed by optional additional visits. The registry will include assessments of various asthma and allergy characteristics to achieve a more flexible, efficient, selective, and inclusive approach to participant recruitment while still following national guidelines to foster participant safety. CAUSE investigators may invite children or adults without asthma or atopic diseases to participate in the registry as "healthy" controls; for validation of laboratory tests, study monitoring equipment, and/or procedures; or for site procedure training of study personnel for certification and quality assurance.

Participants may opt to withdraw their information or discontinue from the registry at any time, in person, by telephone, or in writing.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is either:

   1. At least 18 years old, willing and able to provide informed consent at the time of enrollment
   2. Under the age of 18, accompanied by a legal guardian who is willing and able to provide informed consent at the time of enrollment
2. Participant has a primary place of residence within the Office of Management and Budget (OMB)-defined Metropolitan Statistical Area (MSA)

Exclusion Criteria:

1. Participant does not speak English or Spanish and/or guardian does not speak English or Spanish
2. Participant does not have access to a phone, either personal or public, with regularity that could be used for scheduling and safety follow-up
3. Past or current medical problems or findings from physical examination or laboratory testing, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may affect the quality or interpretation of the data obtained from the study

Participants who are pregnant or lactating will not be excluded or discontinued from the study, but will not undergo any procedures that are prohibited during pregnancy per the Childhood Asthma in Urban Settings 02 (CAUSE-02) Registry for Asthma Characterization and Recruitment 3 (RACR3) Manual of Procedures (MOP)(e.g., allergen skin testing, spirometry) during the pregnancy.

Potential participants may be reassessed as outlined in the Protocol CAUSE-02 MOP.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population enrolled in this registry will be participants living within the Metropolitan Statistical Area (MSA) assigned by the Office of Management and Budget (OMB) for a given clinical site.
  The Protocol Childhood Asthma in Urban Settings 02 (CAUSE-02) Registry for Asthma Characterization and Recruitment 3 (RACR3) eligibility criteria are broad to anticipate diverse recruitment needs for current and future CAUSE protocols.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with asthma and allergy characteristics | 7 years
  Characteristics of the participants enrolled in the registry will be assessed on a periodic basis (descriptive summary of diagnosis and parameters associated with the former).

CONTACTS AND LOCATIONS:
Overall Officials: Christine A. Sorkness, RPh, PharmD, Study Chair — University of Wisconsin School of Medicine and Public Health; Division of Allergy & Immunology; Daniel J. Jackson, MD, Study Chair — University of Wisconsin School of Medicine and Public Health; Division of Allergy & Immunology
Locations (7):
- United States (7):
  - Children's Hospital Colorado: Allergy Program, Aurora, Colorado
  - Children's National Medical Center: Inner City Asthma Consortium (ICAC) Clinical Research Site, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago: Division of Allergy and Immunology, Chicago, Illinois
  - Boston Children's Hospital: Department of Immunology, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai: Division of Clinical Immunology, Immunology Institute, New York, New York
  - Columbia University Medical Center: Department of Medicine, Division of Pulmonary, Allergy and Critical Care Medicine, New York, New York
  - Cincinnati Children's Hospital Medical Center: Asthma Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait